CLINICAL TRIAL: NCT01964339
Title: Obesity Hypoventilation Syndrome Prevalence Study
Status: Terminated | Type: Observational
Why Stopped: This study was stopped due to low recruitment.
Sponsor: Philips Respironics (Industry)
Responsible Party: Sponsor
Other Study IDs: HRC-1240-OHSPREV-MS
Record Dates: First submitted 2013-10-14; First posted 2013-10-17 (Estimated); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Obesity Hypoventilation Syndrome
MeSH Terms: conditions — Obesity Hypoventilation Syndrome | interventions — Blood Gas Analysis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- BMI greater than or equal to 30kg/m2 -venous: BMI greater than or equal to 30kg/m2 scheduled for PSG as part of routine clinical care. Participants will undergo blood draw (venous blood gas and metabolic panel) and data collection from PSG study.
  Interventions: Other: BMI greater than or equal to 30kg/m2 scheduled for PSG. Undergo blood draw (venous blood gas and metabolic panel) and data collection from PSG study.
- BMI greater than or equal to 30kg/m2 - arterial: BMI greater than or equal to 30kg/m2 scheduled for PSG as part of routine clinical care. Participants will undergo blood draw (arterial blood gas and metabolic panel) and data collection from PSG study.
  Interventions: Other: BMI greater than or equal to 30kg/m2 scheduled for PSG. Undergo blood draw (arterial blood gas and metabolic panel) and data collection from PSG study.

INTERVENTIONS:
Other: BMI greater than or equal to 30kg/m2 scheduled for PSG. Undergo blood draw (venous blood gas and metabolic panel) and data collection from PSG study. — Venous blood gas, basic metabolic panel, PSG variable data collection.
  Groups: BMI greater than or equal to 30kg/m2 -venous
Other: BMI greater than or equal to 30kg/m2 scheduled for PSG. Undergo blood draw (arterial blood gas and metabolic panel) and data collection from PSG study. — Arterial blood gas, basic metabolic panel, PSG variable data collection
  Groups: BMI greater than or equal to 30kg/m2 - arterial

SUMMARY:
This is an observational study to characterize the prevalence of Obesity Hypoventilation Syndrome in patients referred to the sleep lab.

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to 21 yrs. of age
* Referred to sleep lab for diagnostic PSG, initial titration PSG or split night PSG as routine clinical care
* BMI greater than or equal to 30kg/m2

Exclusion Criteria:

* Acutely ill or medically unstable to participate per PI
* Current positive airway pressure(PAP therapy)users
* Medical History of Chronic Obstructive Pulmonary Disease(COPD)
* Incapable of providing own informed consent
* BMI less than 30kg/m2

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with a BMI greater than or equal to 30kg/m2 scheduled for a routine polysomnograpy (PSG) test. Participants will be recruited from pulmonology clinics or referred to the sleep lab via hospital admissions.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2013-10-09 (Actual); Primary Completion 2014-05-21 (Actual); Study Completion 2014-05-21 (Actual)

PRIMARY OUTCOMES:
Baseline venous blood draw | single blood draw
  The study involves a venipuncture and data collection at the time of sleep study. Data collection will be correlated to blood draw results.

OTHER OUTCOMES:
Standard polysomnography (PSG) variables | once
  Standard PSG variables will be collected post PSG study. Standard variables include total sleep time, sleep efficiency, hypopneas, apneas (obstructive, central, mixed), stages of sleep, oxygen desaturation (minimum and averages during sleep).
Key demographic characteristics will be collected. | once
  Key demographics will be collected including gender, age, height, and weight. Hip, waist and neck measurements will be collected.

CONTACTS AND LOCATIONS:
Locations (1):
- Ochsner Baptist Medical Center, New Orleans, Louisiana, United States